CLINICAL TRIAL: NCT07101081
Title: GYNGHER - HER2 Expression in Gynecological Malignancies: a Brazilian Cohort
Acronym: GYNGHER
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00061
Record Dates: First submitted 2025-07-16; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Gynaecological Cancers
Keywords: Gynaecological cancers; HER-2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Diagnostic Test: HER-2 Test — Samples from patients with gynecological tumors eligible to the study will be retrospectively identified and the paraffin slides will be sent to central laboratory to perform HER2 IHC testing using the automated protocols (Dako and Ventana). Expert pathologists will select primary tumor samples from surgery or excisional biopsies with enough material to perform HER2 testing using both antibodies without exhausting the cancer tissue. The entire cohort will be tested with both Dako HercepTest and Roche Ventana 4B5 antibody using gastric cancer and breast cancer criteria for positivity (3+, 2+ and 1+, 0).

SUMMARY:
Adult patients with gynecologic cancer (endometrial, ovarian, cervical, vulvar and vaginal cancers) treated at Oncoclínicas & CO sites will be enrolled for primary tumor immunohistochemistry (IHC) analysis. When sufficient paraffin tissue is available for biomarker testing, slides will be sent from partner Pathology Labs of the OC Precision Medicine network to Locus Lab (São Paulo) for HER2 staining with automated protocols (Dako HercepTest and Roche Ventana 4B5) and scoring using different criteria (gastric cancer, breast cancer, and endometrial cancer). Primary objective is to describe the prevalence of HER2 high expression (IHC 3+ using Dako HercepTest and gastric cancer scoring criteria) in endometrial, ovarian, and cervical cancers (common gynecological malignancies). Secondary objectives are to describe the prevalence of HER2 high expression (IHC 3+ using Dako HercepTest and gastric cancer scoring criteria) in vulvar and vaginal cancers (rare gynecological malignancies); and to describe the prevalence of different HER2 expression levels (IHC 0, 1+ and 2+ using Dako HercepTest and gastric cancer scoring criteria) across all gynecological malignancies, to describe HER2 expression levels as per endometrial cancer scoring criteria in the endometrial cohort; to describe the association of different histological subtypes of gynecological cancer with HER2 IHC expression levels.

DETAILED DESCRIPTION:
Retrospective molecular epidemiologic study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at sample collection; - Diagnosis of cervical, endometrial, ovarian/peritoneum/uterine tube, vulvar, or vaginal cancers;
* Sufficient paraffin primary tumor tissue for biomarker testing in the OC Precision Medicine Pathology labs.
* Date of diagnosis of gynecological cancer must be from January 2020 to March 2025.
* Patients need to sign informed consent, or waiver of informed consent is granted.

Exclusion Criteria:

* Patients without sufficient paraffin tissue for the proposed biomarker testing.
* Patients whose diagnosis was performed in metastatic lesion.
* Patients with history of exposure to systemic anti-cancer therapies for the gynecological cancer diagnosis before surgery or excisional biopsy of gynecological cancer (information is available in the original histopathology request document stored in the LIMS).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: In total, 350 samples in total (100 cervical cancer, 100 endometrial cancer, 100 ovarian cancer, and 50 vulvar or vaginal cancer).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
HER2 IHC status as per Dako HercepTest and gastric cancer scoring criteria. | Through study completation,an average of 1 year
  To describe the prevalence of HER2 high expression (IHC 3+) in a cohort of patients in Brazil with gynecological cancers (cervical, endometrial and ovarian cancers).

SECONDARY OUTCOMES:
HER2 IHC status as per Dako HercepTest and gastric cancer scoring criteria. | Through study completation,an average of 1 year
  To describe HER2 expression levels (IHC 0, 1+ and 2+) in a cohort of patients in Brazil with gynecological cancers (cervical, endometrial and ovarian, vulvar and vaginal cancers).

CONTACTS AND LOCATIONS:
Overall Officials: Angélica Nogueira Rodrigues, Principal Investigator — Oncoclínicas Precision Medicine
Locations (1):
- Oncoclínicas Precision Medicine, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/